CLINICAL TRIAL: NCT04518748
Title: A Phase 1 Study of Combined Y-90 Selective Internal Radiation Therapy (Y-90 SIRT) and Stereotactic Body Radiation Therapy (SBRT) in Hepatic Malignancy.
Brief Title: Combined Y-90 Selective Internal Radiation Therapy (Y-90 SIRT) and Stereotactic Body Radiation Therapy (SBRT) in Hepatic Malignancy.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2020.052; HUM00181352 (Other: University of Michigan); R01EB022075 (NIH)
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Liver Malignancy
Keywords: Ytrium-90 (Y-90); Selective Internal Radiation Therapy (SIRT); Stereotactic Body Radiation Therapy (SBRT)
MeSH Terms: interventions — Yttrium-90; Radiosurgery; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Y-90 SIRT followed by SBRT (Experimental): Y-90 SIRT followed by SBRT
  Interventions: Drug: Yttrium-90; Device: Selective Internal Radiation Therapy; Radiation: Stereotactic Body Radiation Therapy; Diagnostic Test: PET/CT; Device: Therasphere

INTERVENTIONS:
Drug: Yttrium-90 — Radioactive isotope Y-90 at day 0, administered by selective internal radiation therapy (SIRT)
  Other Names: Y-90
Device: Selective Internal Radiation Therapy — SIRT at day 0, to administer Yttrium-90 (Y-90) Theraspheres
  Other Names: SIRT
Radiation: Stereotactic Body Radiation Therapy — 3-5 fractions over 1-2 weeks, after Y-90 SIRT
  Other Names: SBRT
Diagnostic Test: PET/CT — Within 3 hours of completing Y-90 SIRT
Device: Therasphere — Glass microspheres containing Y-90, administered at day 0 by SIRT

SUMMARY:
This study will investigate the combination of Ytrium-90 (Y-90) Selective Internal Radiation Therapy (SIRT) followed by Stereotactic Body Radiation Therapy (SBRT). Y-90 SIRT alone or SBRT alone are standard procedures used in the treatment of liver cancer. This study will assess the combination of Y-90 SIRT and SBRT and obtain preliminary information about the side effects and safety of the combination therapy. Additionally, this is the first time that Y-90 PET-CT imaging will be included in planning for SBRT.

DETAILED DESCRIPTION:
Selective Internal Radiation Therapy (SIRT) is a technique where radiation is internally delivered to a tumor. In SIRT, small radioactive beads are deposited in the liver through a large blood vessel (hepatic artery). SIRT that uses the radioactive material Yttrium-90 is called Y-90 SIRT.

Stereotactic Body Radiation Therapy (SBRT) is a technique where radiation is externally delivered to a tumor. In SBRT, a machine produces a beam of radiation that targets the tumor from outside the body.

After receiving Y-90 SIRT, participants will be evaluated to estimate how much radiation was absorbed by their tumors during Y-90 SIRT. Y-90 PET-CT imaging will be used to help plan SBRT, which will target areas of tumors that did not receive as much radiation as expected during Y-90 SIRT.

Updated to add 5 patients to enrollment goal to achieve desired number of evaluable patients

Since patients treated with Y-90 for any liver malignancy can benefit from the Y-90+SBRT combined treatment approach we have decided to open up the protocol to all eligible patients and not HCC alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unresectable hepatocellular carcinoma or metastatic liver cancer. Hepatocellular carcinoma is defined as having at least one of the following:

  * Biopsy proven hepatocellular carcinoma (HCC); or
  * A discrete hepatic tumor(s) as defined by the Barcelona imaging criteria.

Metastatic liver cancer is defined as having:

o pathological confirmation of any metastatic disease with a new or enlarging liver lesion consistent with metastases. The targeted lesion does not need to be biopsied if the patient has a known history of metastatic disease

* Patients must not have known untreated or progressive disease outside of the liver
* At least one lesion >2 cm diameter or 4 cc volume
* Patients must have a life expectancy of at least 6 months.
* Patients must be 18 years of age or older
* All men, as well as women of childbearing potential, must agree to use effective contraception throughout the study and for 90 days following treatment.
* Patients must understand and be willing to sign an informed consent form approved for this purpose by the Institutional Review Board (IRB) of the University of Michigan Medical Center indicating that they are aware of the investigational aspects of the treatment and the potential risks.

Exclusion Criteria:

* Inability to lie still for imaging studies (e.g. PET/CT)
* Pregnancy or nursing females or refusal to use birth control in patients capable of reproduction.
* Patients with known allergy or contraindication to intravenous iodinated contrast agents
* Patients with an allergy or contraindication to MRI on MRI contrast (Eovist or Gadolinium)
* Contraindication to Theraspheres

  * Tc-99m macroaggregated albumin (MAA) hepatic arterial perfusion scintigraphy showing any deposition to the gastrointestinal tract that may not be corrected by angiographic techniques
  * Shunting of blood to the lungs that could result in delivery of greater than 30 Gy to the lungs.
  * Hepatic artery catheterization contraindication; such as patients with vascular abnormalities or bleeding diathesis;
  * Bilirubin >2.0 at baseline
  * Occlusion of the main portal vein
* Contraindication to radiation therapy
* Note: Patients who have an increase in bilirubin >1.0 from the time of Y90 to SBRT or his/her bilirubin goes above 2.5 after Y90 will not be eligible for SBRT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change in Child-Turcotte-Pugh (CTP) score >= 2 points from baseline | Up to 6 months after SBRT
  The primary safety endpoint is the binary indicator for a CTP increase of 2 or more points within 6 months and relative to pre-SBRT baseline. An increase of 2 or more points indicates clinically significant liver decompensation.
Incidence of toxicities of grade 3 or higher | Up to 6 months after SBRT
  A secondary safety endpoint is grade 3+ toxicity within 6 months relative to pre-SBRT baseline. Assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of patients with a change in albumin + bilirubin (ALBI) level of >= 0.5 | Up to 6 months after SBRT
  A secondary safety endpoint is the binary indicator for an increase in ALBI within 6 months relative to pre-SBRT baseline of 0.5 or greater.

SECONDARY OUTCOMES:
Freedom from local progression (FFLP) at the lesion level | Until progression or last surveillance scan at approximately 24 months after SBRT
  FFLP at the lesion level is defined as the time from SIRT to progression of a SBRT-treated lesion. Progression is defined based on RECIST and mRECIST criteria.
Freedom from local progression (FFLP) at patient level | Until progression or last surveillance scan at approximately 24 months after SBRT
  FFLP at the patient level is defined as the time from SIRT to progression of the treated lesions including those not targeted by SBRT. Progression is defined based on RECIST v1.1and mRECIST criteria.
Response rate | Up to 6 months after SBRT
  Response rate defined per RECIST v1.1 and mRECIST criteria and categorized as follows: progressive disease or stable disease = non-responder, partial response or complete response = responder.
Overall survival | Until death from any cause, or until patient's last follow-up visit, or until study stops; up to approximately 5 years.
  Overall survival will be calculated as the time from Y-90 SIRT treatment to death from any cause, or until patient's last follow-up visit, or until study stops.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Cuneo, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No